CLINICAL TRIAL: NCT01480882
Title: "A Prospective, Cross-over Randomized Trial to Assess the Efficacy and Safety of Mechanical Percussor "LEGA" Compared With Conventional Chest Physiotherapy in Adults With Chronic Bronchiectasis or Chronic Obstructive Pulmonary Disease (COPD
Brief Title: Efficacy and Safety Study of a Percussion Device to Mobilise Sputum From Respiratory Passage
Acronym: LEGA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Penang Hospital, Malaysia (Other Government)
Responsible Party: Principal Investigator, Dr.Ong Loke Meng, Head, Clinical Research Centre, Penang Hospital, Malaysia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CT-11-HPP-001; NMRR-11-661-10072 (Registry Identifier: National Medical Reseach Register (NMRR))
Record Dates: First submitted 2011-11-20; First posted 2011-11-29 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Bronchiectasis; Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Manual percussion; Mechanical percussion; Chronic bronchiectasis; Chronic Obstructive Pulmonary Disease; Wet sputum weight; Dry sputum weight
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Chest PhysioTherapy (Active Comparator): Conventional Chest Physiotherapy (CCPT) is delivered by professional physiotherapist for 15 minutes.
  Interventions: Procedure: Conventional Chest Physiotherapy (CCPT)
- Mechanical percussion (Experimental): Mechanical percussion will be delivered by a device called "LEGA" for 15 minutes
  Interventions: Device: Mechanical percussion (LEGA)

INTERVENTIONS:
Procedure: Conventional Chest Physiotherapy (CCPT) — Conventional chest percussion will be applied for a duration of 15 minutes.
  Other Names: Manual percussion
  Arms: Conventional Chest PhysioTherapy
Device: Mechanical percussion (LEGA) — Mechanical chest percussion will be delivered by a device for 15 minutes.
  Other Names: LEGA
  Arms: Mechanical percussion

SUMMARY:
A Malaysian company by name Formedic Technologies SDN BHD has devised a hand held machine which is supposed to mimic the chest percussion performed by professional physiotherapist to mobilize sputum through the respiratory passage.

The aim of this study is to compare the effectiveness and safety of this mechanical percussion device in the treatment of airway clearance with conventional chest physiotherapy carried out by qualified physiotherapists in patients suffering from bronchiectasis or Chronic obstructive Pulmonary disease (COPD).

DETAILED DESCRIPTION:
This study will compare the amount of sputum expectorated during the two procedures and not intended to look at the clinical improvement of the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients > 18 years of age
2. Chronic sputum expectoration-(producing >30ml/day of sputum at baseline)
3. Clinical diagnosis of bronchiectasis or COPD
4. Not carrying out regular chest physiotherapy (for the purposes of this study this will be defined as less than two occasions per week)
5. Clinically stable disease (defined as no requirement for antibiotics in the 4 weeks preceding study entry).
6. FEV1 of > 35% of the predicted value in COPD patients

Exclusion Criteria:

1. Primary diagnosis of asthma;
2. Active sarcoidosis
3. Active Pulmonary tuberculosis.
4. History of brittle bones,
5. History of broken ribs in the past one year.
6. History of severe osteoporosis
7. Bleeding from the lungs or haemoptysis
8. Experiencing intense pain in the thoracic region
9. Clinical suspicion of increased intracranial pressure.
10. Have head or neck injuries
11. Have collapsed lungs or a damaged chest wall;
12. Recent myocardial infarction, unstable angina and stroke (Within 6 months prior to enrollment)
13. Have a pulmonary embolism or lung abscess;
14. Have an active hemorrhage
15. Have injuries to the spine
16. Have open wounds or burns in the thoracic region
17. Have had recent surgery (Within six months prior to enrollment.)
18. Any systemic steroids within 4/52 prior to enrollment
19. Any antibiotics within 4/52 prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Comparing the 'wet weight' and 'dry weight' of the sputum expectorated during 20 minutes of the two procedures. | 6 days
  The patients will be instructed to cough out the sputum into a preweighed container during the 15 minutes of the procedure(Manual or mechanical percussion)and 5 minutes after the procedure.Container will be weighed to get the wet weight of the sputum then will be dried in a laboratory oven at 60degree c for 48 hours and weighed again to get the dry weight of the sputum

SECONDARY OUTCOMES:
Change in FEV1 and FVC before and after the two methods of therapy | 15 minutes after completion of the procedure compared to baseline
  Any changes in the lung function will be measured as - FEV1 (%predicted) and FVC (%predicted)
Changes in pulse, blood pressure and respiratory rate | 15 minutes after completion of treatment compared to baseline
  Monitoring of Pulse, blood pressure, respiratory rate, skin colour and patients reaction to treatment.
Patient preference | After completing 6 days of participation in the study
  Patients will be participating in the study for 6 days. On the 6th day after completion of treatment they will be required to answer a simple questionnaire to find out if they prefer one procedure over the other and why.

CONTACTS AND LOCATIONS:
Overall Officials: Ong L Meng, MBBS, FRCP, Study Chair — Penang Hospital, Malaysia; Mohd I Izmi, MBBS, MD, Principal Investigator — Penang Hospital, Malaysia
Locations (1):
- Penang hospital, George Town, Pulau Pinang, Malaysia

REFERENCES:
- See also: Click here for more information about this study- NMRR-11-661-10072 — http://www.nmrr.gov.my